CLINICAL TRIAL: NCT07112183
Title: An Open Label Study to Assess Efficacy of Oral Treprostinil Titrated to 3.0mg Three Times Daily or Highest Tolerable Dose in 30 Patients With Symptomatic Primary or Secondary Raynaud's Phenomenon Resistant to Standard Vasodilatory Therapy
Brief Title: Open Label Treprostinil Raynaud's Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Aaron Waxman MD PhD, Executive Director, Center for Pulmonary Heart Diseases, Director, Pulmonary Vascular Disease Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001219
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Raynaud's Disease; Raynaud Phenomena; Raynauds
Keywords: Raynaud's; Raynaud's Disease; Raynaud's Phenomena; Connective Tissue Disease; Systemic Sclerosis
MeSH Terms: conditions — Raynaud Disease; Connective Tissue Diseases; Scleroderma, Systemic | interventions — treprostinil

STUDY DESIGN:
Intervention Model Description: 30 patients with symptomatic primary or secondary Raynaud's phenomenon (RP) resistant to standard vasodilatory therapy will be enrolled. Prior to treatment, subjects will record each day for 42 days the number of RP attacks as well as the duration of each RP attack, considered to be baseline data. After the 6-week baseline run in, all subjects will receive oral treprostinil sustained release tablets. Dose escalations can occur every 48 hours in 0.125 mg increments. Subjects will be titrated as tolerated to a goal dose of 3mg three times daily over a 6-week period. Titration can be done as quickly as tolerated. Once at goal dose subjects will enter the 26-week treatment phase. Throughout the study (6-week titration - 26-week treatment phase) subjects will record each day the number of RP attacks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- An open label study to assess efficacy of oral treprostinil in patients with Raynaud's (Experimental): A single center open label study to assess efficacy of oral treprostinil titrated to a tolerable goal dose of 3.0 mg three times per day (TID) in 30 patients with symptomatic primary or secondary Raynaud's phenomenon resistant to standard vasodilatory therapy. Eligible subjects at the time of signing an informed consent will have a diagnosis of primary or secondary Raynaud's phenomenon. Once enrolled, subjects will enter a run in period and record each day for 42 days the number of RP attacks as well as the duration of each RP attack. Frequency and duration of RP recorded within 6-weeks before active treatment phase will be baseline data. After the run in period subjects will be titrated as tolerated to a goal dose of 3mg TID over a 6-week period. Throughout the study (6-week titration - 26-week treatment phase) subjects will record each day the number of RP attacks as well as the duration of each RP attack.
  Interventions: Drug: Oral treprostinil (UT-15C) sustained release tablets

INTERVENTIONS:
Drug: Oral treprostinil (UT-15C) sustained release tablets — 30 patients with symptomatic primary or secondary Raynaud's phenomenon (RP) resistant to standard vasodilatory therapy will be enrolled. Prior to treatment, subjects will record each day for 42 days the number of RP attacks as well as the duration of each RP attack, considered to be baseline data. After the 6-week baseline run in, all subjects will receive oral treprostinil sustained release tablets. Dose escalations can occur every 48 hours in 0.125 mg increments. Subjects will be titrated as tolerated to a goal dose of 3mg three times daily over a 6-week period. Titration can be done as quickly as tolerated. Once at goal dose subjects will enter the 26-week treatment phase. Throughout the study (6-week titration - 26-week treatment phase) subjects will record each day the number of RP attacks.

SUMMARY:
Raynaud's phenomenon is a condition where the blood vessels in participants fingers and toes get too narrow when cold or stressed. This makes participants fingers and toes change colors - they might turn white, then blue, and finally red as blood flow returns. It can be painful and cause numbness or tingling.

When participants have Raynaud's, blood vessels react too strongly to cold or stress. Fingers and toes may turn white (blood moves away from the area), blue (lack of oxygen), or red and feel painful or tingly when warming up. These episodes usually last from a few minutes to several hours.

There are two types of Raynaud's. Primary Raynaud's (also called Raynaud's disease) itself and isn't connected to other health problems. It's the most common type and affects mostly women under 30. Secondary Raynaud's (also called Raynaud's phenomenon) is caused by other diseases like lupus, scleroderma, or rheumatoid arthritis. This type tends to be more serious and may cause painful sores on fingertips called digital ulcers.

For mild cases, staying warm might be enough. But if symptoms are severe, participants doctor might prescribe various medications including calcium channel blockers - blood pressure medicines that help open blood vessels, or other vasodilators - medicines that widen blood vessels. About 40% of people with scleroderma develop painful sores on their fingertips called digital ulcers. These happen when there isn't enough blood flow to heal small injuries.

For severe cases with digital ulcers, doctors might use prostacyclin therapy - medicines that mimic a natural substance that opens blood vessels. Oral treprostinil is a newer pill form of prostacyclin therapy that helps improve blood flow. The investigators are conducting a research study testing whether oral treprostinil - a pill that mimics prostacyclin (a natural blood vessel opener) - can help people with severe Raynaud's that doesn't respond to usual treatments. This represents hope for better treatment options for people with the most challenging cases of this condition.

ELIGIBILITY:
Inclusion Criteria:•

* Patients aged ≥ 18 years
* Active Raynaud's Phenomenon defined as patients with refractory RP having four or more RP attacks per week in the 4 weeks before inclusion in the study despite stable background vasodilator treatment for at least 3 months.
* Patients with primary Raynaud's Phenomenon
* Patients with Raynaud's secondary to connective tissue diseases (including scleroderma (SSc), limited scleroderma (CREST), mixed connective tissue disease (MCTD), primary Sjogren's syndrome (SS), systemic lupus erythematosus (SLE), with diagnosis of the underlying rheumatic disease based on standard criteria.
* Patients on stable dose phosphodiesterase inhibitors (sildenafil, tadalafil or vardenafil), endothelin antagonists, alpha adrenergic antagonists, or calcium channel blockers defined as 3-months with no change in dose will be allowed to participate.

Exclusion Criteria:

* Uncontrolled hypertension, diabetes mellitus, acute coronary or cerebrovascular event within 3 months, evidence of malignancy, history of sympathectomy
* Smoking within 3 months or smoking cessation using nicotine products
* Subjects with history of diverticulosis
* Subjects with moderate to severe liver disease, Child Pugh Class B or C
* Subjects currently taking any other prostacyclin.
* Pregnant or breast feeding or considering pregnancy in next 4 months
* Participation in trial with an investigational drug within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Raynaud's Condition Score from baseline (6-week run in), comparing treprostinil treatment phase vs. baseline phase. | 38 weeks
  Once enrolled, throughout the study (6-weeks before active treatment; 6-week titration; 26-week treatment phase) subjects will record each day the number of RP attacks as well as the duration of each RP attack.. Frequency and duration of RP recorded within 6-weeks before active treatment phase will be considered to be baseline data.
  Every day subjects will complete the Raynaud's Condition Score (RCS). The RCS is an 11-point numerical rating scale (0-10) where 0 = "no difficulty" and 10 = "extreme difficulty". Patients complete the scale daily, and the average scores are calculated. The scale asks patients to consider multiple factors when rating their difficulty, including the number and duration of Raynaud's attacks, symptoms such as pain, numbness, burning, and tingling, and how the condition affects their ability to use their hands and perform daily activities.

SECONDARY OUTCOMES:
Digital Ulcer Score | 32 Weeks
  Digital Ulcer Score (DUS) will be assessed at every 4-week visit, Weeks 4, 8, 12, 16, 20, 24 and 28. Minimum Value: 0; No theoretical maximum. Higher scores indicate worse outcomes (more severe digital ulcers). The DUS is calculated by assessing each individual ulcer and multiplying the depth of the ulcer (1 point for hyperkeratosis, 10 points for ulcer) by the diameter (1 point if <0.5 cm, 2 points for ≥0.5 cm). The total score is then calculated as the sum of all individual ulcer scores.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron B Waxman, MD, PhD, Principal Investigator — Brigham and Women's Hospital, Pulmonary Vascular Disease Program
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Maverakis E, Patel F, Kronenberg DG, Chung L, Fiorentino D, Allanore Y, Guiducci S, Hesselstrand R, Hummers LK, Duong C, Kahaleh B, Macgregor A, Matucci-Cerinic M, Wollheim FA, Mayes MD, Gershwin ME. International consensus criteria for the diagnosis of Raynaud's phenomenon. J Autoimmun. 2014 Feb-Mar;48-49:60-5. doi: 10.1016/j.jaut.2014.01.020. Epub 2014 Feb 1. PMID 24491823
- [Background] Shah AA, Schiopu E, Hummers LK, Wade M, Phillips K, Anderson C, Wise R, Boin F, Seibold JR, Wigley F, Rollins KD. Open label study of escalating doses of oral treprostinil diethanolamine in patients with systemic sclerosis and digital ischemia: pharmacokinetics and correlation with digital perfusion. Arthritis Res Ther. 2013 Apr 18;15(2):R54. doi: 10.1186/ar4216. PMID 23597147
- [Background] Milio G, Corrado E, Genova C, Amato C, Raimondi F, Almasio PL, Novo S. Iloprost treatment in patients with Raynaud's phenomenon secondary to systemic sclerosis and the quality of life: a new therapeutic protocol. Rheumatology (Oxford). 2006 Aug;45(8):999-1004. doi: 10.1093/rheumatology/kel038. Epub 2006 Feb 16. PMID 16484290
- [Background] Roustit M, Blaise S, Allanore Y, Carpentier PH, Caglayan E, Cracowski JL. Phosphodiesterase-5 inhibitors for the treatment of secondary Raynaud's phenomenon: systematic review and meta-analysis of randomised trials. Ann Rheum Dis. 2013 Oct;72(10):1696-9. doi: 10.1136/annrheumdis-2012-202836. Epub 2013 Feb 20. PMID 23426043
- [Background] Denton CP, Hachulla E, Riemekasten G, Schwarting A, Frenoux JM, Frey A, Le Brun FO, Herrick AL; Raynaud Study Investigators. Efficacy and Safety of Selexipag in Adults With Raynaud's Phenomenon Secondary to Systemic Sclerosis: A Randomized, Placebo-Controlled, Phase II Study. Arthritis Rheumatol. 2017 Dec;69(12):2370-2379. doi: 10.1002/art.40242. PMID 29193819
- [Background] Garcia de la Pena Lefebvre P, Nishishinya MB, Pereda CA, Loza E, Sifuentes Giraldo WA, Roman Ivorra JA, Carreira P, Rua-Figueroa I, Pego-Reigosa JM, Munoz-Fernandez S. Efficacy of Raynaud's phenomenon and digital ulcer pharmacological treatment in systemic sclerosis patients: a systematic literature review. Rheumatol Int. 2015 Sep;35(9):1447-59. doi: 10.1007/s00296-015-3241-1. Epub 2015 Apr 1. PMID 25824427
- [Background] Costa E, Cunha-Santos F, Dourado E, Oliveira D, Falzon L, Romao V, Duarte AC, Cordeiro A, Santiago T, Sepriano A. Systematic literature review to inform the Portuguese recommendations for the management of Raynaud's phenomenon and digital ulcers in systemic sclerosis and other connective tissue diseases. ARP Rheumatol. 2024 Jul 1;3(Apr-Jun):128-144. doi: 10.63032/YHBL8967. PMID 38306796
- [Background] Khouri C, Lepelley M, Bailly S, Blaise S, Herrick AL, Matucci-Cerinic M, Allanore Y, Trinquart L, Cracowski JL, Roustit M. Comparative efficacy and safety of treatments for secondary Raynaud's phenomenon: a systematic review and network meta-analysis of randomised trials. Lancet Rheumatol. 2019 Dec;1(4):e237-e246. doi: 10.1016/S2665-9913(19)30079-7. PMID 38229380
- [Background] Flavahan NA, Flavahan S, Mitra S, Chotani MA. The vasculopathy of Raynaud's phenomenon and scleroderma. Rheum Dis Clin North Am. 2003 May;29(2):275-91, vi. doi: 10.1016/s0889-857x(03)00021-8. PMID 12841295
- [Background] Stjernbrandt A, Pettersson H, Lundstrom R, Liljelind I, Nilsson T, Wahlstrom J. Incidence, remission, and persistence of Raynaud's phenomenon in the general population of northern Sweden: a prospective study. BMC Rheumatol. 2022 Jul 21;6(1):41. doi: 10.1186/s41927-022-00272-0. PMID 35858907
- [Background] Maciejewska M, Sikora M, Maciejewski C, Alda-Malicka R, Czuwara J, Rudnicka L. Raynaud's Phenomenon with Focus on Systemic Sclerosis. J Clin Med. 2022 Apr 28;11(9):2490. doi: 10.3390/jcm11092490. PMID 35566614
- [Background] Curtiss P, Svigos K, Schwager Z, Lo Sicco K, Franks AG Jr. Part I: Epidemiology, pathophysiology, and clinical considerations of primary and secondary Raynaud's phenomenon. J Am Acad Dermatol. 2024 Feb;90(2):223-234. doi: 10.1016/j.jaad.2022.06.1199. Epub 2022 Jul 7. PMID 35809798